CLINICAL TRIAL: NCT06550076
Title: A Phase 3, Multicenter, Open-Label Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of TAK-279 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of TAK-279 in Participants With Moderate-to-Severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-279-PsO-3003; 2024-512496-12-00 (EU CTIS Number); jRCT2031240413 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis
Keywords: Latitude Psoriasis 3; Latitude Research Program; Latitude PsO OLE

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A (De Novo Cohort) + Part B (Open Label Extension): TAK-279 (Experimental): Part A: Participants will receive TAK-279, oral tablet once daily (QD) for up to 52 weeks.
  Part B: Participants who completed the treatment period of parent studies (TAK-279-3001 [NCT06088043], TAK-279-3002 [NCT06108544], or TAK-279-PsO-3004 [NCT06973291]) or who completed Part A will receive TAK-279, oral tablet QD for up to 156 weeks.
  Interventions: Drug: TAK-279

INTERVENTIONS:
Drug: TAK-279 — TAK-279 oral tablet

SUMMARY:
The main aim of this study is to check the side effects of TAK-279 and how well it is tolerated in participants with moderate-to-severe plaque psoriasis.

All participants will be assigned to study treatments of TAK-279 and will be treated with TAK-279 if the participants meet the study rules.

Participants will be in the study for up to 217 weeks, including up to 35 days for the screening period, 52 weeks (Part A) up to 156 additional weeks (Part B) study treatment and 4 weeks follow up period. During the study, participants will visit their study clinic multiple times.

DETAILED DESCRIPTION:
This study consists of 2 parts: Part A and Part B.

Part A: Participants who did not participate in one of the parent studies (TAK-279-3001 [NCT06088043], TAK-279-3002 [NCT06108544], or TAK-279-PsO-3004 [NCT06973291]) may be enrolled and will be treated for up to 52 weeks. Participants who successfully complete Part A of the study are eligible to continue in Part B, but investigators must confirm their eligibility to continue in Part B.

Part B: Participants who complete the treatment period of TAK-279-3001 (NCT06088043), TAK-279-3002 (NCT06108544), or TAK-279-PsO-3004 (NCT06973291) parent studies or who complete Part A are eligible to enroll directly into open label extension treatment in Part B and will be treated for up to 156 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

Part A:

* Participant is willing and able to understand and fully comply with study procedures and requirements (including digital tools and applications), in the opinion of the investigator.
* Participant has provided written informed consent and any required privacy authorization before the initiation of any study procedures.
* Participant is aged 18 years or older at the time of consent.
* Participant has a diagnosis of chronic plaque psoriasis for >=6 months prior to the screening visit.
* Participant has stable plaque psoriasis defined as no significant flare or change in morphology (as assessed by the investigator) in psoriasis for >=6 months before screening.
* Participant has moderate-to-severe plaque psoriasis as defined by a PASI score >=12 and a sPGA score >=3 at screening and Day 1.
* Participant has plaque psoriasis covering >=10% of his or her total BSA at screening and Day 1.
* Participant must be a candidate for phototherapy or systemic therapy.

Part B:

- Participant has completed 52 weeks of treatment (TAK-279-3001 or Part A) or 60 weeks of treatment (TAK-279-3002), or 16 weeks of treatment (TAK-279-PsO-3004) in their parent study.

Main Exclusion Criteria

Part A:

* Participant has evidence of non-plaque psoriasis (erythrodermic, pustular, predominantly guttate psoriasis, predominantly inverse, or drug-induced psoriasis). If a participant meets criteria for inclusion based on typical plaque psoriasis presentation, a limited amount of inverse psoriasis is not exclusionary.
* Participant requires systemic treatment, other than nonsteroidal anti-inflammatory drugs, during the trial period for an immune-related disease (e.g., inflammatory bowel disease).
* Participant has any clinically significant medical condition, evidence of an unstable clinical condition (e.g., cardiovascular, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, or immunologic), or vital signs/physical/laboratory/ECG abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of study results. These include but are not limited to:

  1. Participant has a history of known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
  2. Participant had a major surgery within 60 days prior to Day 1 or has a major surgery planned during the study.
  3. Participant has unstable, poorly controlled, or severe hypertension at screening, confirmed by 2 repeat assessments.
  4. Participant has a history of Class III or IV congestive heart failure as defined by New York Heart Association criteria.
  5. Participant has a history of cancer or lymphoproliferative disease, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
  6. For participants with asthma, chronic obstructive pulmonary disease, or other pulmonary illnesses, participant has been hospitalized in the past 3 months, has ever required intubation for treatment, currently requires oral corticosteroids, or has required more than 1 course of oral corticosteroids within 6 months prior to Day 1.
  7. Participant has any of the following cardiovascular disease history: A new diagnosis of atrial fibrillation or an episode of atrial fibrillation with rapid ventricular response or other dysrhythmia, non-acute cardiac hospitalization (e.g., pacemaker implantation), pulmonary embolism, or deep venous thrombosis within the past 6 months prior to screening. Any history of cerebrovascular event, myocardial infarction, coronary stenting, or aortocoronary bypass surgery. If, however, the investigator determines there are no suitable treatment alternatives available for the participant and it has been at least 6 months since the occurrence of any such event, the participant may enroll.
  8. Participant has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if he or she participated in the study, in the opinion of the investigator.
  9. Participant has significant/uncontrolled psychiatric illness, in the opinion of the investigator.
  10. Participant has any lifetime history of suicidal ideation, suicidal behavior, or suicidal attempts by 1) medical history; or 2) by Columbia-Suicide Severity Rating Scale (C-SSRS) documentation at screening or by answering "yes" to Question 5 for suicidal ideation on the C-SSRS at screening; or 3) is clinically deemed to have a suicide risk by the investigator.
  11. Participant has a patient health questionnaire - 8 (PHQ-8) score of 15 or above at screening.
  12. Participant has a history of clinically significant drug or alcohol abuse within 12 months prior to Day 1.
* Participant has received any of the following biologics or biosimilar versions within the time frame indicated or 5 half-lives, whichever is longer:

  1. Antibodies to interleukin (IL) -12/-23, IL-17, or IL-23 (eg, ustekinumab, secukinumab, tildrakizumab, ixekizumab, or guselkumab) within 6 months prior to Day 1.
  2. Tumor necrosis factor inhibitor(s) (e.g., etanercept, adalimumab, infliximab, certolizumab) within 2 months prior to Day 1.
  3. Agents that modulate integrin pathways to impact lymphocyte trafficking (e.g., natalizumab) or agents that modulate B cells or T cells (e.g., alemtuzumab, abatacept, or visilizumab) within 3 months prior to Day 1.
  4. Rituximab or other immune cell-depleting therapy within 6 months prior to Day 1.
* Participant has any previous exposure to TAK-279 (also known as NDI-034858) or other TYK2 inhibitors, including deucravacitinib, or participant participated in any study that included a TYK2 inhibitor (e.g., deucravacitinib, VTX958, GLPG3667, etc.), unless the participant has documentation of post-trial unblinding that confirms the partcipant did not receive a TYK2 inhibitor.
* Participant has a known or suspected allergy to TAK-279 or any of its components.

Part B:

* Participant has completed the parent study or Part A but was permanently discontinued from treatment.
* Participant had evidence of significant noncompliance with study visits or study drug in the parent study or Part A, as defined in the parent study protocol or in the opinion of the investigator.
* Participant has met criteria for termination from the parent study or Part A, regardless of whether or not the participant was terminated from the parent study or Part A.
* Participant has developed evidence of non-plaque psoriasis (erythrodermic, pustular, predominantly guttate psoriasis, predominantly inverse, or drug-induced psoriasis) since enrollment in the parent study or Part A.
* Participant has developed a concomitant comorbid skin condition that, in the opinion of the investigator, would interfere with the study assessments.
* Participant has received a prohibited psoriasis treatment during the parent study or Part A, whether or not that treatment was documented as a concomitant medication and is expected to continue that treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1950 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAE) | From start of the drug administration up to Week 56 (Part A) and Week 160 (Part B)
  A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. An SAE is any untoward medical occurrence that at any dose: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event in the opinion of the healthcare provider, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. TEAEs consist of both serious and non-serious adverse events.

SECONDARY OUTCOMES:
Part A and B: Number of Participants Achieving 75% Improvement from Baseline in Psoriasis Area and Severity Index (PASI-75) Score | Baseline up to Week 52 (Part A) and Week 156 (Part B)
  The PASI is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. The PASI-75 is defined as 75% improvement from baseline in PASI score.
Part A and B: Number of Participants Achieving a Static Physician's Global Assessment (sPGA) of Clear (0) or Almost Clear (1) With a >=2-point Decrease from Baseline | Baseline up to Week 52 (Part A) and Week 156 (Part B)
  The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean greater than (>) 0, less than (<) 1.5; Mild (2) = mean greater than or equal to (>=) 1.5, <2.5; Moderate (3) = mean >=2.5, <3.5; and Severe (4) = mean >=3.5.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (278):
- United States (74):
  - Total Dermatology, Birmingham, Alabama
  - University of Alabama Hospital - Whitaker Clinic -, Birmingham, Alabama
  - Cahaba Dermatology Skin Health Center, Hoover, Alabama
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Saguaro Dermatology Associates, LLC - Probity - PPDS, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Johnson Dermatology Clinic, Fort Smith, Arkansas
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Zenith Research, Inc., Beverly Hills, California
  - First OC Dermatology Research Inc., Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Long Beach Research Institute, Long Beach, California
  - Metropolis Dermatology Downtown LA - Probity - PPDS, Los Angeles, California
  - UCLA University of California Los Angeles, Los Angeles, California
  - Northridge Clinical Trials, Northridge, California
  - UC Davis Dermatology Clinic, Sacramento, California
  - TCR Medical Corporation, San Diego, California
  - University Clinical Trials, San Diego, California
  - Dermatology Institute and Skin Care Center, Santa Monica, California
  - UNISON Clinical Trials (Shahram Jacobs md inc.), Sherman Oaks, California
  - Driven Research LLC, Coral Gables, Florida
  - Revival Research Corporation - Florida - ClinEdge - PPDS, Doral, Florida
  - FXM Clinical Research Ft. Lauderdale, LLC, Fort Lauderdale, Florida
  - Direct Helpers Medical Center, Hialeah, Florida
  - Florida Academic Centers Research, Miami, Florida
  - FXM Clinical Research Miami, LLC, Miami, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - FXM Research Miramar, Miramar, Florida
  - Renstar Medical Research -21 NE 1st Ave, Ocala, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Advanced Clinical Research Institute (ACRI) - Florida, Tampa, Florida
  - Divine Dermatology and Aesthetics, LLC, Atlanta, Georgia
  - Marietta Dermatology & The Skin Cancer Center - Marietta, Marietta, Georgia
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - Georgia Skin and Cancer Clinic, Savannah, Georgia
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Arlington Dermatology, Rolling Meadows, Illinois
  - NorthShore Medical Group Dermatology - Skokie, Skokie, Illinois
  - DS Research - 1005 E. Lewis & Clark Pkwy Indiana Location, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Dermatology Specialists Research - 3810 Springhurst Blvd, Louisville, Kentucky
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - University of Michigan Hospital - 1500 E Medical Center Dr, Ann Arbor, Michigan
  - Oakland Hills Dermatology - 3400 Auburn Rd, Auburn Hills, Michigan
  - Revival Research Corporation - ClinEdge, Troy, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Skin Specialists PC, Omaha, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - Dartmouth Hitchcock Medical Center - Old Etna Rd, Lebanon, New Hampshire
  - ALLCUTIS Research, LLC., Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Sadick Research Group, New York, New York
  - Montefiore AOA - BRANY, The Bronx, New York
  - Accellacare of Cary, Cary, North Carolina
  - The Skin Surgery Center for Clinical Research - Objective Health - PPDS, Winston-Salem, North Carolina
  - Bexley Dermatology Research - Probity - PPDS, Bexley, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Oregon Medical Research Center PC, Portland, Oregon
  - University of Pittsburgh Medical Center-3601 5th Ave, Pittsburgh, Pennsylvania
  - Cumberland Skin Center for Clinical Research - Objective Health - PPDS, Hermitage, Tennessee
  - International Clinical Research US LLC, Murfreesboro, Tennessee
  - Arlington Research Center, Arlington, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - UT Physicians Dermatology - Bellaire Station, Bellaire, Texas
  - Modern Research Associates, Dallas, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - San Antonio, San Antonio, Texas
  - Texas Dermatology and Laser Specialists-San Antonio-7703 Floyd Curl Dr, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Houston Center for Clinical Research, LLC, Sugar Land, Texas
  - Center For Clinical Studies, LTD. LLP - 451 N Texas Ave, Webster, Texas
  - Virginia Clinical Research - 6160 Kempsville Cir, Norfolk, Virginia
- Argentina (3):
  - Conexa Investigación Clínica S.A., Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro de Investigaciones Médicas Tucumán, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigacion Clinica, Ciudad Autónomade Buenos Aires
- Australia (5):
  - St George Dermatology and Skin Cancer Center - Probity - PPDS, Kogarah, New South Wales
  - The Skin Center - Probity, Benowa, Queensland
  - Skin Health Institute Inc - Probity - PPDS, Carlton, Victoria
  - Alfred Health, Parkville, Victoria
  - Western Health - Sunshine Hospital, Parkville, Victoria
- Bulgaria (11):
  - Medical Center Unimed EOOD-Sevlievo, Sevlievo, Gabrovo
  - Medical Center Asklepii OOD, Dupnitsa, Kyustendil
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Sofia-Grad
  - Diagnostic Consultative Centre - Focus-5 - LZIP EOOD, Sofia, Sofia-Grad
  - Medical Center Hera EOOD-Sofia, Sofia, Sofia-Grad
  - Diagnostic Consultative Center XXVIII - Sofia - EOOD, Sofia, Sofia-Grad
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - MC Comac Medical, Sofia, Sofia-Grad
  - Multiprofile Hospital For Active Treatment Dr Tota Venkova, Gabrovo
  - Diagnostic Consultative Center Sveti, Haskovo
  - Medical Center Medconsult Pleven OOD, Pleven
- Canada (31):
  - Beacon Dermatology - Probity, Calgary, Alberta
  - Dermatology Research Institute, Inc., Calgary, Alberta
  - Alberta DermaSurgery Centre - Probity, Edmonton, Alberta
  - VIDA Dermatology - Probity, Edmonton, Alberta
  - Care Clinic, Red Deer, Alberta
  - Enverus Medical Research - Probity, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Karma Clinical Trials, St. John's, Newfoundland and Labrador
  - CCA Medical Research - Probity, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre - Probity, Barrie, Ontario
  - Kingsway Clinical Research - Probity, Etobicoke, Ontario
  - Guelph Dermatology Research - Probity, Guelph, Ontario
  - Lima's Excellence In Allergy And Dermatology Research (Leader) Inc. - Probity, Hamilton, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Mediprobe Research Inc, London, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc - Probity, Markham, Ontario
  - DermEdge Research - Probity, Mississauga, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation | Newmarket, Canada, Newmarket, Ontario
  - North Bay Dermatology Center - Probity, North Bay, Ontario
  - The Centre for Clinical Trials Inc., Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre For Dermatology, Richmond Hill, Ontario
  - North York Research Inc. - Probity, Toronto, Ontario
  - Canadian Dermatology Centre - Probity, Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Toronto Research Centre - Probity, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Siena Medical Research Corporation, Montreal, Quebec
  - Skinsense Medical Research - Probity, Saskatoon, Saskatchewan
- China (25):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology (HUST), Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Huashan Hospital Fudan University - PPDS, Shanghai, Minhang District
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - The 2nd Hospital of Xi'An Jiaotong University, Xi'an, Shan'xi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The 1st Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
- Czechia (10):
  - Dermamedica, s.r.o. - Kozni Ambulance Nachod, Náchod, Královéhradecký kraj
  - Nemocnice AGEL Novy Jicin a.s, Nový Jičín, Moravskoslezský kraj
  - CCR Ostrava s.r.o., Ostrava, Moravskoslezský kraj
  - Dermskin s.r.o, Olomouc, Olomoucký kraj
  - Pratia Pardubice a.s. - PRATIA - PPDS, Pardubice, Pardubický kraj
  - Pratia Brno s.r.o. - PRATIA - PPDS, Brno, South Moravian
  - CLINTRIAL s.r.o., Prague
  - Prof. MUDr. Petr Arenberger, DrSc. - CRC - PPDS, Prague
  - Praglandia, Prague
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- France (4):
  - Office of Mireille Ruer-Mulard, MD, Martigues, Paca
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - Hopital Charles Nicolle-1 Rue de Germont, Rouen
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
- Germany (7):
  - Hautarztpraxis Mahlow, Blankenfelde-Mahlow, Brandenburg
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Klinikum Oldenburg, Oldenburg, Lower Saxony
  - Klinische Forschung Dresden Gmbh, Dresden, Saxony
  - Praxis fur Dermatologie and Venerologie, Dresden, Saxony
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - Dermatologikum Hamburg, Hamburg
- Hungary (4):
  - Allergo-Derm Bakos Kft., Szolnok, Jász-Nagykun-Szolnok
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Markusovszky Egyetemi Oktatókórház, Szombathely, Vas County
  - Debreceni Egyetem, Debrecen
- Israel (2):
  - Rabin Medical Center - PPDS, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (3):
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Presidio Ospedaliero Gaspare Rodolico, Catania, Sicily
  - Azienda Usl Toscana Centro - Firenze, Florence, Tuscany
- Japan (17):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hino Dermatology Clinic, Fukutsu-shi, Fukuoka
  - Takagi Dermatological Clinic, Obihiro-Shi, Hokkaidô
  - JR Sapporo Hospital, Sapporo, Hokkaidô
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaidô
  - Fukuoka University Hospital, Fukuoka, Hukuoka
  - Nippon Life Hospital, Osaka, Osaka
  - Seikoukai Omi Medical Center, Kusatsu-shi, Shiga
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Tokyo Teishin Hospital, Sumida-Ku, Tokyo
  - Medical Corporation Jitai-kai Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo-To
  - Shirasaki Dermatology Clinic, Takaoka-shi, Toyama
  - Ohyama Dermatology Clinic, Kumamoto
  - Tokyo Medical University Hospital, Tokyo
  - Dermatology and Ophthalmology Kume Clinic, Sakaishi, Ôsaka
- Latvia (8):
  - Smite Aija medical practice in dermatology, venerology, Talsi, Talsu Aprinkis
  - Semigallia, Kuldīga
  - Riga 1st Hospital, Riga
  - Aesthetic dermatology clinic of prof. J. Kisis, Riga
  - Health Center 4-1 Grebenscikova Str, Riga
  - Veseliba un estetika Ltd., Riga
  - Outpatient Clinic Adoria, Riga
  - Health Center 4-Skanstes iela 50, Riga
- Poland (49):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Twoja Przychodnia PCM, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne ALL-MED, Krakow, Lesser Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Katowice - PRATIA, Katowice, Lower Silesian Voivodeship
  - Globe Badania Kliniczne Spolka z o.o. - Klodzko, Kłodzko, Lower Silesian Voivodeship
  - Cityclinic Przychodnia lekarsko psychologiczna Matusiak sp.p, Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions Sp. z o.o. S.K., Lublin, Lublin Voivodeship
  - Luxderm Specjalistyczny Gabinet Dermatologiczny Dorota Krasowska, Lublin, Lublin Voivodeship
  - Centrum Terapii Współczesnej J.M. Jasnorzewska S.K.A., Lódz, Lódzkie
  - Rheumatology Clinic NZOZ Lecznica MAK-MED, Nadarzyn, Masovian Voivodeship
  - ETG Siedlce - PPDS, Siedlce, Masovian Voivodeship
  - RCMed Oddzial Sochaczew, Sochaczew, Masovian Voivodeship
  - Clinical Best Solutions Sp. z o.o. S.K., Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Clinical Research Group Sp. z o.o, Warsaw, Masovian Voivodeship
  - High-Med Przychodnia Specjalistyczna, Warsaw, Masovian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - ETG Warszawa - PPDS, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Dermatologia, Warsaw, Masovian Voivodeship
  - FutureMeds - Targowek - PPDS, Warsaw, Masovian Voivodeship
  - NZOZ Osteo Medic SC Artur Racewicz Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Spolka Komandytowa, Bialystok, Podlaskie Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o, Szpital Sw. Wojciecha, Oddzial Dermatologii, Gdansk, Pomeranian Voivodeship
  - Centrum Badan Klinicznych Pi-house Sp. Z O. O., Gdansk, Pomeranian Voivodeship
  - Derm-art, Gdynia, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Silesian Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - Twoja Przychodnia Szczecińskie Centrum Medyczne Sp. z o.o., Szczecin, West Pomeranian Voivodeship
  - Centrum Uslug Medycznych MaxMed, Bochnia
  - Centrum Medyczne Bydgoszcz- PRATIA, Bydgoszcz
  - Ambulatorium Sp. z o.o., Elblag
  - Promed P. Lach R. Głowacki Sp. j., Centrum Medyczne Promed, Krakow
  - Diamond Clinic Sp. z o.o., Diamond Medical Center, Krakow
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Lodzi, Klinika Dermatologii i Wenerologii, Lodz
  - Pro Life Medica Sp. z o.o. ETG Lublin, Lublin
  - Twoja Przychodnia - Nowosolskie Centrum Medyczne sp. z o.o, Nowa Sól
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - MICS Centrum Medyczne Torun, Torun
  - Royalderm Agnieszka Nawrocka, Warsaw
  - dermMEDICA Sp. z o.o. | Krzysztofa Kolumba 6, Wroclaw
  - Dermoklinika-Centrum Medyczne s.c, Lodz, Łódź Voivodeship
  - Velocity Skierniewice Sp. z o.o., Skierniewice, Łódź Voivodeship
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
  - Ostrowieckie Centrum Medyczne Anna Olech Cudzik Krzysztof Cudzik s.c., Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- GCM Medical Group, San Juan, Puerto Rico
- South Korea (10):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Chosun University Hospital, Gwangju, Gwangju Gwang'yeogsi
  - Seoul National University Bundang Hospital, Beon-gil Bundang-gu, Gyeonggi-do
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggido
  - Konkuk University Medical Center, Gwangjin-Gu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seocho-Gu, Seoul Teugbyeolsi
  - Soon Chun Hyang University Hospital Seoul, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (2):
  - Hospital Clinico San Carlos, Donostia / San Sebastian, Guipúzcoa
  - Hospital de Manises, Manises, Valencia
- Taiwan (6):
  - National Cheng Kung University, Tainan, Tainan City
  - National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Mackay Memorial Hospital-Taipei branch, Taipei
  - National Taiwan University Hospital, Zhong Zheng Qu
- United Kingdom (6):
  - Velocity Clinical Research - High Wycombe - PPDS, High Wycombe, Buckinghamshire
  - 4 Medical Clinical Solutions - Swinton - PPDS, Ilford, Essex
  - Salford Royal Hospital - PPDS, Salford, Lancashire
  - Whipps Cross University Hospital, London, London, City of
  - Accellacare of Northamptonshire, Harrow, Middlesex
  - Velocity Clinical Research North London - Percy Road - PPDS, London, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed — https://clinicaltrials.takeda.com/study-detail/7c0533db1af5404d